CLINICAL TRIAL: NCT04122885
Title: Study of Plasma Tumor-promoting Factors and Immune Function After Explorative Laparotomy, Tumor Debulking and HIPEC (Hyperthermic Intraperitoneal Chemotherapy) vs. PIPAC (Pressurized IntraPeritoneal Aerosol Chemothereapy) in Patients With Peritoneal Metastasis as Evaluated by Serum Proliferative Activity, Levels of Proteins, Cytokines, Circulating Growth Factors, Inhibitors and Their Binding Proteins.
Brief Title: Study of Plasma Tumor-promoting Factors and Immune Function After Laparotomy, Cytoreductive Surgery and HIPEC vs. PIPAC in Patients With Peritoneal Metastasis
Acronym: IMMUNOPAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 392/2018BO1
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Peritoneal Cancer; Chemotherapy-Induced Change
Keywords: HIPEC; PIPAC; cytoreductive surgery; immune function; cytokines; plasma proteins
MeSH Terms: interventions — Oxaliplatin; Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRS and HIPEC: Cyroreductive surgery and Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
  Interventions: Procedure: Cytoreductive surgery and Hyperthermic IntraPeritoneal Chemotherapy
- PIPAC: Pressurized IntraPeritoneal Aerosol Chemotherapy (if CRS and HIPEC not possible)
  Interventions: Combination Product: PIPAC with oxaliplatin

INTERVENTIONS:
Combination Product: PIPAC with oxaliplatin — Oxaliplatin 92 mg/m2 BSA, applied as an aerosol for 30 min under normothermic conditions at 12-15 mmHg pressure
  Groups: PIPAC
Procedure: Cytoreductive surgery and Hyperthermic IntraPeritoneal Chemotherapy — If complete cytoreduction possible (CC-0). Application time 60 min, T 41-43 °C
  Other Names: CRS and HIPEC
  Groups: CRS and HIPEC

SUMMARY:
The general goal of this study is to investigate the effect of treatment on serum concentrations of proteins known to impact angiogenesis or tumor growth and establishment in patients with peritoneal metastasis of various origin. Since the immune system is thought, by many, to have an impact on tumor growth and development, this study also seeks to determine the impact of abdominal surgery on postoperative immune function in PM patients, as judged by proteins known to influence immune function. This study will not only characterize the postoperative plasma but also to determine if the magnitude of any of the changes noted is associated with a worse or improved oncologic outcome.

The principle purpose of this study is to gather perioperative serum/plasma samples from patients with PM from a variety of different primary tumors (ovarian, gastric, and colorectal) undergoing either CRS and HIPEC versus PIPAC.

DETAILED DESCRIPTION:
The plasma samples obtained in this protocol will also be used to study the various plasma proteins that influence immune function as well as those that influence angiogenesis. In addition to the proteins mentioned above, there are also a large number of other proteins that have not been investigated thus far in the perioperative window; these proteins also merit assessment. The plasma obtained via this study and protocol will also be used to search for other tumor growth factors influenced by surgery or to investigate the impact of surgery on immune function.

Aim 1: To determine perioperative serum levels, over time, of a variety of serum proteins including but not limited to IGFBP-3, VEGF, Ang 2, PlGF, sVCAM, CHI3L1, MMP-2, MMP-3, MCP-1 and proteins that influence immune function as well as other proteins in the following 2 groups of patients:

1. PM patients treated with CRS and HIPEC
2. PM patients treated with PIPAC.

Aim 2: To compare the perioperative blood protein results between the 2 different groups of patients.

Aim 3: To determine, within each group, a possible correlation between the magnitude of these effects on oncological outcome (patient overall survival).

Aim 4: To search for other surgery-influenced plasma or cellular factors that may influence early postoperative tumor growth or that hold promise as tumor or prognostic markers.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (18 years of age or older) with ovarian, gastric, or colorectal cancer who have PM who after thorough evaluation are deemed candidates for:

* CRS & HIPEC if complete cytoreductive surgery is possible (OR)
* PIPAC if no complete cytoreductive surgery is possible at the University Hospital of Tubingen are eligible for entry in this study

Exclusion Criteria:

* ASA 3 & 4 patients
* Patients who have received chemotherapy within 1 month prior to the planned surgery
* Patients who have received blood transfusion(s) within 2 weeks of the planned surgery
* Patients in whom the treatment plan includes systemic chemotherapy to be given during the first 2 weeks after surgery.
* History of allergic reaction to cisplatin or other platinum containing compounds or doxorubicin
* Severe renal impairment, myelosuppression, severe hepatic impairment, severe myocardial insufficiency, recent myocardial infarction, severe arrhythmias
* Immunocompromised patients such as those taking an immunosuppressive medication and those who have a known disease of the immune system
* Patients or family members involved in the planning and conduct of the study (applies to University of Tübingen staff involved)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the institutions involved. All patients must meet inclusion/exclusion criteria (as indicated above) to be considered.
  Each subject will undergo medical examination during the screening visit (Visit 1) prior to enrolment. The personal data and detailed medical history will be recorded. The screening will take place no more than 6 weeks before intervention. This screening procedure will consist of:
  * Checking of inclusion/exclusion criteria
  * Detailed history including medical history
  * A standard physical examination including the cardiovascular, nervous, respiratory systems, conscience, memory, orientation, and body weight
  The patient's informed consent for study participation will be signed at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum levels of the proteins of interest over time | 6 weeks

SECONDARY OUTCOMES:
Postoperative complications | 30 days
Overall survival | 18 months
  Measured from time point of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Reymond, MD MBA, Principal Investigator — National Center for Pleura and Peritoneum
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
IPD might be shared on request after completion of the study

REFERENCES:
- See also: University Hospital Tübingen — https://www.medizin.uni-tuebingen.de/en-de/startseite